CLINICAL TRIAL: NCT06929078
Title: Role of Individualized Positive End-expiratory Pressure Versus Fixed Positive End-expiratory Pressure in Mechanical Ventilation During Laparoscopic Surgeries
Brief Title: Role of Individualized PEEP Vs Fixed PEEP in Mechanical Ventilation During Laparoscopic Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Noor-Ul-Ain (Other)
Responsible Party: Sponsor-Investigator, Noor-Ul-Ain, Post Graduate Resident Anesthesiology Fellowship of College of Physicians and Surgeons Pakistan, Combined Military Hospital Bahawalpur
Organization: Combined Military Hospital Bahawalpur (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HospitalBahawalpur
Record Dates: First submitted 2025-03-27; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Laparoscopic Surgery; Pneumoperitoneum; Positive End Expiratory Pressure (PEEP)
Keywords: mechanical ventilation; lung compliance; positive end-expiratory pressure; respiratory mechanics; oxygenation index; driving pressure
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5cm of water Positive End-expiratory Pressure will be applied after induction of general anesthesia (Placebo Comparator): A fixed positive end-expiratory pressure of 5cm of water will administered to the participants after induction of general anesthesia during mechanical ventilation undergoing laparoscopic surgeries.
  Interventions: Other: Protective lung ventilation methods with different positive end-expiratory pressure during Laparoscopic Surgeries
- Individualized PEEP with recruitment maneuver guided by driving pressure measurement (Experimental): Recruitment maneuver will be applied after induction of general anesthesia and indiviualized positive end-expiratory pressure will be applied guided by driving pressue during mechanical ventilation during laparoscopic surgeries.
  Interventions: Other: Protective lung ventilation methods with different positive end-expiratory pressure during Laparoscopic Surgeries
- Conventional ventilation (No Intervention): Conventional ventilation method without additional positive end-expiratory pressure will be applied to participants during mechanical ventilation undergoing laparoscopic surgeries.

INTERVENTIONS:
Other: Protective lung ventilation methods with different positive end-expiratory pressure during Laparoscopic Surgeries — Protective lung ventilation methods with positive end-expiratory pressure help in prevention of atelectasis and improvement of intraoperative ventilator parameters e.g low driving pressure and improved dynamic compliance resulting in better oxygenation of lungs ere will be three groups in this study. Individualized positive end-expiratory pressure with recruitment maneuver and fixed positive end-expiratory pressure will be interventional groups. They will be compared with conventional ventilation group in which no additional positive end-expiratory pressure will be applied. The effects on respiratory parameters and oxygenation of patients will be compared for each group. This study will determine which method of positive end-expiratory pressure is superior and how it differs from conventional ventilation for prevention of atelectasis induced by pneumoperitonium and improvement of respiratory mechanical parameters and oxygenation in Mechanical ventilation during laparoscopic surgeries.
  Other Names: Application of possitive end expiratory pressure during laparoscopic surgeries; Individual PEEP with recruitment maneuver; Fixed PEEP; Protective lung ventilation; Different positive end-expiratory pressure strategies
  Arms: 5cm of water Positive End-expiratory Pressure will be applied after induction of general anesthesia; Individualized PEEP with recruitment maneuver guided by driving pressure measurement

SUMMARY:
To compare the effects of Individualized positive end-expiratory pressure with recruitment maneuver on respiratory parameters and oxygenation in mechanical ventilation during laparoscopic surgeries with the fixed positive end-expiratory pressure and conventional mechanical ventilation without positive end-expiratory pressure.

DETAILED DESCRIPTION:
Thus study will compare the effects different methods of positive end-expiratory pressure administration in mechanical ventilation on respiratory parameters and oxygenation of the patients undergoing laparoscopic surgeries. There will be three groups of patients which will be as follows: Individualized positive end-expiratory pressure with recruitment maneuver group, fixed positive end-expiratory pressure group and conventional mechanical ventilation. Respiratory parameters; dynamic compliance, driving pressure and ratio of partial pressure of oxygen to fractional inspiration of oxygen will be measured. Mechanical ventilation respiratory parameters i .e. peak pressure, plateu pressure , dynamic compliance and driving pressure will be measured from ventilator machine. P/F ratio( Ratio of partial pressure of oxygen to inspiratory fraction of oxygen) will be measured by taking blood samples for arterial blood gas analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age Limit : 25 years to 65 years

  2. Patients undergoing laparoscopic suregeries

  3. ASA 1-3

Exclusion Criteria:

* 1. Hemodynamic instability 2. Bronchospam 3. Patients having COPD 4. History of pulmonary bulla 5. Patients having history of pneumothora

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Driving pressure | 10 minutes after induction of general anesthesia, 10 minutes after pneumoperitonium creation and 10 minutes before extubation of patient
  Driving pressure is defined as airway plateau pressure minus positive end-expiratory pressure and reflects the degree of ventilator induced trauma. Airway plateau pressure and positive end-expiratory values will be taken from ventilator monitor.
Dynamic compliance of lungs | 10 minutes after induction of general anesthesia, 10 minutes after pneumoperitonium creation and 10 minutes before extubation of patient
  Dynamic compliance is change in lung volume by the change in pressure in the presence of airflow and is calculated by dividing tidal volume of a breath with difference between peak pressure of airway and positive end-expiratory pressure. Tidal volume, peak airway pressure and positive end-expiratory pressure will be noted from ventilator machine monitor.
Oxygenation Index | 10 minutes after induction of general anesthesia and 10 minutes before extubation of patient
  Oxygenation index is calculated by following formula:
  OI = Mean Airway Pressure × FiO2 × 100 ÷ PaO2 FiO2 (fractional inspiration of oxygen) and PaO2 (partial pressure of oxygen) will be recorded from arterial blood gas analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Colonal Naseem Abbas, Principal Investigator — Head of Department of Anesthesia Combined Military Hospital Bahawalpur; Dr Noor-Ul-Ain Registrar Anesthesia, Principal Investigator — Department of Anesthesia Combined Military Hospital Bahawalpur
Locations (1):
- Combined Military Hospital Bahawalpur, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez-Bustamante A, Sprung J, Parker RA, Bartels K, Weingarten TN, Kosour C, Thompson BT, Vidal Melo MF. Individualized PEEP to optimise respiratory mechanics during abdominal surgery: a pilot randomised controlled trial. Br J Anaesth. 2020 Sep;125(3):383-392. doi: 10.1016/j.bja.2020.06.030. Epub 2020 Jul 16. PMID 32682559
- [Background] Simon P, Girrbach F, Petroff D, Schliewe N, Hempel G, Lange M, Bluth T, Gama de Abreu M, Beda A, Schultz MJ, Pelosi P, Reske AW, Wrigge H; PROBESE Investigators of the Protective Ventilation Network* and the Clinical Trial Network of the European Society of Anesthesiology. Individualized versus Fixed Positive End-expiratory Pressure for Intraoperative Mechanical Ventilation in Obese Patients: A Secondary Analysis. Anesthesiology. 2021 Jun 1;134(6):887-900. doi: 10.1097/ALN.0000000000003762. PMID 33843980